CLINICAL TRIAL: NCT02910128
Title: Childhood Obesity Prevention Trough the "CHIQUICHEFS" Program of Education Innovation and Cooking in a Primary School: A Quasi Experimental Study
Brief Title: Childhood Obesity Prevention Trough Education Innovation in Primary School: A Quasi-experimental Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital El Escorial (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2
Record Dates: First submitted 2016-09-05; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Childhood Obesity; Dietary Habits; Quality of Life
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- School intervention (Experimental): chiquichefs education innovation
  Interventions: Behavioral: chiquichefs
- control school (No Intervention): A primary schools will function as control schools.

INTERVENTIONS:
Behavioral: chiquichefs — A project based learning using healthy trough cooking as the core of the curriculum, so children learn the academic content through cooking workshop of mediterranean diet in their school.
  Arms: School intervention

SUMMARY:
This study evaluates the effect of the education innovation program"chiquichefs" on anthropometric variables, quality of life and nutritional habits in an elementary school children. Compared with a control group of the same age but in another school.

DETAILED DESCRIPTION:
Childhood obesity is recognized as both the most prevalent health problem in the western world and as a global epidemic. It has an multifactorial aetiology. Obesity in children has been attributed to decrease in physical activity and the overconsumption of cheap energy dense food.

Spain has one of the highest prevalence rates of overweight and obese children among OECD countries.

Health promotion and prevention strategies in community settings are in general most effective where they engage with social networks and build social capital to enable community ownership and embedding strategies. This is particularly the case for health promotion at primary school, as social institutions within a community setting that represent a complex system with direct an indirect community relationship and social networks.

One of the best methods to prevent childhood obesity is to follow the Mediterranean diet. Especially in Mediterranean countries for the ease of access to essential products of this diet.

Chiquichefs is a methodology of project-based learning using healthy through cooking as the core of the curriculum, so children learn the academic content through cooking workshop in their school.

A quasi-experimental study was developed, for which children of the intervention schools (n = 75) in a public spanish school is compared with children of a control schools (n = 75) in the same region.

The interventions started in october 2015. In the intervention school, a whole-school approach named "chiquichefs" is implemented with the aim of improving culinary skills and dietary behaviour.

The "chiquichefs" project ideas is to make the kitchen the central pillar of the curriculum for several years. So children will learn to cook during school hours -- and not as an after-school activity -- and along the way they will also be taught the core content.

They'll do maths counting chick peas, study the recipes of literature, the geography of food, work out the boiling point of soups and learn the anatomy of cattle.

With this project, we aim to deliver the core educational requirements, teach kids to cook and lay the foundations for them to benefit from a healthier diet throughout their lives. We're going conduct a scientific study to measure the impact on the children's health and education in the hope of eventually persuading others to follow our lead.

We are going to measure the anthropometric variables, the adherence to mediterranean diet and the quality of life of all participants before and after the "chiquichefs" program.

ELIGIBILITY:
Inclusion Criteria:

* All children and their caregivers enrolled at the participating schools and that agree to sign informed consent.

Exclusion Criteria:

* None except not agreement to sign the informed consent.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Child absolute change in BMI Z-score, based on weight and height | 1 year
  Weight is measured using a weighing scale, to the nearest 0.1 kg; height is measured using a measuring rod, to the nearest 0.1 cm. These two measurements are used to calculate the BMI, BMI was compared this with the graphics BMI standardized for Spanish population ( kg/m2).

SECONDARY OUTCOMES:
Adherence to mediterranean diet | 1 year
  kidmed index questionnaire at the beginning and end of the project
Quality of life | 1 year
  kidscreen-10 questionnaire at the beginning and end of the project

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willeboordse M, Jansen MW, van den Heijkant SN, Simons A, Winkens B, de Groot RH, Bartelink N, Kremers SP, van Assema P, Savelberg HH, de Neubourg E, Borghans L, Schils T, Coppens KM, Dietvorst R, Ten Hoopen R, Coomans F, Klosse S, Conjaerts MH, Oosterhoff M, Joore MA, Ferreira I, Muris P, Bosma H, Toppenberg HL, van Schayck CP. The Healthy Primary School of the Future: study protocol of a quasi-experimental study. BMC Public Health. 2016 Jul 26;16:639. doi: 10.1186/s12889-016-3301-9. PMID 27456845
- [Result] Foster GD, Sherman S, Borradaile KE, Grundy KM, Vander Veur SS, Nachmani J, Karpyn A, Kumanyika S, Shults J. A policy-based school intervention to prevent overweight and obesity. Pediatrics. 2008 Apr;121(4):e794-802. doi: 10.1542/peds.2007-1365. PMID 18381508
- See also: short documentary video ( spanish) — https://www.youtube.com/watch?v=_KfqcBnqmPE